CLINICAL TRIAL: NCT06616298
Title: Improving Person-Centered Outcomes for Older Adults With Cancer Discharged to Skilled Nursing Facilities and Their Family Caregivers
Brief Title: ALIGN for Older Adults With Cancer in SNFs
Acronym: ALIGN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 24-0548.cc; K23AG076866 (NIH)
Record Dates: First submitted 2024-09-12; First posted 2024-09-27 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Advanced Cancer
Keywords: Skilled Nursing Facility; Caregiver
MeSH Terms: interventions — Health Services Needs and Demand

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Older patients with advanced cancer (Experimental): Older adults with advanced cancer from the University of Colorado Hospital being discharged to skilled nursing facilities (SNF).
  Interventions: Other: Assessing and Listening to Individual Goals and Needs (ALIGN)
- Caregivers of older patients with advanced cancer (Experimental): Caregivers of older adults with advanced cancer from the University of Colorado Hospital being discharged to skilled nursing facilities.
  Interventions: Other: Assessing and Listening to Individual Goals and Needs (ALIGN)
- Control Arm (No Intervention): Control arm participants will receive enhanced usual care. Patients will be provided resources for advance care planning and interact with SNF staff and involved providers who may refer them to palliative care or hospice like previous rigorous palliative care trials.

INTERVENTIONS:
Other: Assessing and Listening to Individual Goals and Needs (ALIGN) — Assessing and Listening to Individual Goals and Needs (ALIGN). ALIGN utilizes the skills of palliative care social workers (PCSWs) trained in family and systems-level theory to address changing preferences for care, family distress, and to facilitate communication across care transitions to improve care aligned with preferences. A patient navigator supports the patient/caregiver and social worker dynamic by helping patients access care and resources. The intervention is implemented virtually in community SNFs and follows patients for 45 days after SNF discharge to reflect real-world patient flow.
  Arms: Caregivers of older patients with advanced cancer; Older patients with advanced cancer

SUMMARY:
The goal of this clinical trial is to learn if it is possible to deliver a palliative care intervention called ALIGN (Assessing and Listening to Individual Goals and Needs) to hospitalized older adults with advanced cancer who are discharged to a skilled nursing facility and their caregivers. The main questions it aims to answer are:

* Can the investigator successfully deliver the ALIGN intervention in different skilled community nursing facilities?
* Can the investigator successfully collect information from participants throughout the study?
* How can the investigator best prepare caregivers to make medical decisions for loved ones that become unable to do so themselves?

Researchers will compare ALIGN to care as it is usually delivered.

Participants will:

* Visit virtually with an ALIGN palliative care social worker every 1-2 weeks during their skilled nursing facility stay and up to 45 days after discharge from the facility or will see a palliative care clinician if recommended by their oncologist or other involved clinician.
* Participants will provide information about how they are doing 1 month, 3 months, and 6 months after enrolling in the study.

ELIGIBILITY:
Patients

Inclusion Criteria:

1. Adults between 18-98 years
2. Stage II-IV solid tumors
3. Discharging from an acute care hospital to a SNF in Colorado
4. English speaking
5. Receiving or establishing care at the University of Colorado Cancer Center
6. If a patient lacks capacity, a legal surrogate decision-maker will be approached to provide proxy consent.
7. Must have access to the technology needed to complete consenting visit and subsequent intervention visits. This includes internet access through a computer, tablet, or smartphone OR cellular service with adequate allowance of cellular minutes to allow virtual visits (by participant's assessment).

Exclusion Criteria:

1. Discharging with hospice care
2. Age less than 18
3. Lacking capacity without a legal surrogate decision maker or proxy. Patient with limited English

Caregivers

Inclusion Criteria:

1. Patient-selected
2. Age ≥ 18
3. English speaking
4. Able to complete baseline measures.

Exclusion Criteria:

1. Discharging with hospice care
2. Age < 18
3. Caregivers with limited English proficiency will be excluded as ALIGN intervention content and documents have only been validated in an English-speaking population.

SNF Staff

Inclusion Criteria:

1. One of 25 interdisciplinary clinicians from the 5 most common community SNFs
2. Staff must be employed by on of the 5 most common community SNFs named above. (care managers, social workers, nurses, physical therapists, occupational therapists, advanced practice providers, and physicians)

Exclusion Criteria:

1. Not employed by one of the top 5 community SNFs patients were discharged to during the pilot trial

PCSW

Inclusion Criteria:

1. PCSWs who conducted the ALIGN intervention and consent to an interview

Ages: 18 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-08-24 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Intervention fidelity as assessed by fidelity checklist | 2.5 years
  Intervention fidelity will be assessed using a fidelity checklist. ALIGN will be considered feasible if there is ≥ 80% adherence to the fidelity checklist for the initial visit, ≥ 80 of at least 1 intervention domain delivered in follow up visits, and if a discharge note is entered for enrolled patients.
Intervention fidelity as assessed by audio-recordings | 2.5 years
  Intervention visits will be recorded and a qualitative analysis will be completed to provide an indepth understanding of fidelity to the core intervention components of ALIGN.
Assessment of treatment contamination in community skilled nursing facilities | 2.5 years
  The investigators will determine the proportion (% total) of caregivers in the control arm who reported that they received components of the ALIGN intervention during the skilled nursing facility stay. ALIGN will be considered feasible if contamination where ALIGN effects usual care is less than 10%.
The proportion (% total) of screened patients that are eligible for enrollment in the trial | 2.5 years
  The investigators will determine the proportion of screened patients (% total) who meet the inclusion criteria
The proportion (% total) of enrolled patients that are assessed for patient-centered outcomes | 2.5 years
  The investigators will determine the proportion of (% total) of enrolled patients that are succesfully assessed for patient-reported and patient-centered outcomes (please see secondary outcomes below)
The proportion (% total) of enrolled caregivers that are assessed for person-centered outcomes | 2.5 years
  The investigators will determine the proportion of (% total) of enrolled caregivers that are succesfully assessed for person-centered outcomes (please see secondary outcomes below)
The proportion (% total) of enrolled patients that are randomized | 2.5 years
  The investigators will determine the proportion of (% total) of enrolled patients that are succesfully randomized
The proportion (% total) of enrolled caregivers that are randomized | 2.5 years
  The investigators will determine the proportion of (% total) of enrolled caregivers that are succesfully randomized

SECONDARY OUTCOMES:
Assessing changes in days at home | 6 months after randomization
  In this exploratory outcome measure, days at home will be calculated as 180 days minus the number of inpatient days in an acute care facility, an inpatient rehabilitation facility, a skilled nursing facility, or an inpatient hospice unit.
Assessing Changes in hospice length of stay | 6 months after randomization
  In this exploratory outcome measures, changes in the length of a hospice stay in both arms of the clinical trial will be measured
Health Care Utilization | 6 months after randomization
  Rehospitalization and emergency department visits for any cause and receipt of chemotherapy within 14 days of death will be collected
Change in quality of life as assessed by the Functional Assessment of Chronic Illness Therapy - Palliative Care (FACIT-PAL-14) | At enrollment and then at 1, 3, and 6 months after randomization
  In this exploratory outcome measure, patients will be asked to complete this 14 item Likert-type scale that measures four primary quality of life domains: physical well-being, social/family well-being, emotional well-being, functional well-being, and spiritual well-being. Scores range from 0-56. Lower scores indicate lower quality of life.
Changes in agreement with health-related outcome statements as assessed by the Attitude Scale | From enrollment and then 1, 3 and 6 months after randomization
  In this exploratory outcome measure, patients will be asked to complete the Attitude Scale which is a 5-point Likert scale that identifies the extent to which patients agree with 8 health-related outcome statements such as: The most important thing to me is living as long as I can, no matter what my quality of life is. Changes in agreement will be measured in both groups of the trial.
Change in frailty as assessed by the Practical Geriatric Assessment | From enrollment and then 1, 3, and 6 months after randomization
  In this exploratory outcome measure, patients and caregivers will be asked to complete this 19 item assessment measures individual domain impairments in areas of physical function, nutrition/weight loss, social support, psychological, comorbidities, and cognitive functioning to guide treatment decisions. There is no composite score for this measure, rather scores from each domain help identify impairments. Higher scores in the physical function, comorbidities, psychological health, domain suggest greater impairment. Lower scores in cognitive and nutritional domains suggest greater impairment.
Change in Advance Care Planning Documentation | From enrollment and then at 6 months after randomization
  Advance Care Planning documents such as Medical Durable Power of Attorney (MDPOA) forms, cardiopulmonary resuscitation (CPR) directives, and the Medical Orders for Scope of Treatment (MOST) forms are documents that communicate end of life wishes for patients and also who they would designate to make medical decisions on their behalf if they are unable to do so themselves. We are measuring completion rates and changes to wishes expressed in these documents in all patients who participate in the trial.
Changes in the Perception of Patient Centeredness of Care Delivered as assessed by the Perception of Patient Centeredness of Care Measure | At enrollment and then 1, 3, and 6 months after randomization
  In this exploratory outcome measure, patients and caregivers will be asked to complete this 18-item instrument using a 4-point Likert scale. Scores range from 18 -72. Higher scores indicate a greater perception of patient-centeredness of care.
Changes in caregiver coping as assessed by the Brief-Cope Questionaire | At enrollment and 1, 3, and 6 months after randomization
  This scale ascertains how people are responding emotionally to a serious circumstance and will be completed by caregivers in this study as an exploratory outcome measure. Scores are presented over three overarching coping styles (problem-focused, emotion-focused, and avoidant) as average scores indicating the degree to which the respondent has been engaging in that coping style. Scores for each coping strategy can range from 2-8. We will measure changes in coping styles over the course of the trial.
Changes in illness understanding and coping support as assessed by the Advanced Illness Coordinating Care Survey | At enrollment and then 1, 3, and 6 months after randomization
  In this exploratory outcome measure, this 5 question survey assesses perceived illness understanding and coping support. The range of scores is from 0 - 24 with higher scores indicating increased illness understanding and coping support.
Changes in the experience of feeling heard and understood as assessed by the Heard and Understood Survey | At enrollment and then 1, 3, and 6 months after randomization
  In this exploratory outcome measure, this 4 question Likert scale survey will be completed by patients and caregivers to assess how well they felt heard and understood by their oncology team of clinicians. Scores can range from 0-16. Higher scores indicate delivery of higher quality care.
Change in the burden or benefits of caregiving as assessed by the Caregiver Reaction Assessment | At enrollment and then at 1, 3 and 6 months after randomization
  In this exploratory outcome measure, caregivers will be asked to complete this 24 item instrument designed to measure the reactions of family members to caring for adults with a variety of illness. The instrument focuses on five dimensions: caregiver esteem, lack of family support, impact on finances, impact on schedule, and impact on health. The minimum score is 0 and the maximum score is 24. A higher score indicates greater caregiver burden.
Changes in congruence between patient and oncologist understanding of the goals of treatment | At enrollment and then post-intervention protocol completion
  In this exploratory outcome measure, patients, caregivers, and oncologists will be asked a focus of treatment question (Please select one of the options below that best describes your current focus of treatment) and asked to select from the following options: curative, life prolonging/rehabilitative, or comfort focused. Patients, caregivers, and oncologists will be asked this question at enrollment and when patients are discharged from ALIGN after the protocol has been completed. We are measuring whether there is increased congruence in the response between patient and their oncologists.
Assessing Oncology Clinican Acceptability | After completion of the ALIGN protocol
  Involved oncology clinicians will be asked using a Likert scale survey their experience working with the ALIGN social worker conducting the intervention in this exploratory outcome measure.
Assessing the Bereaved Caregivers Satisfaction with Care During the Last Month of Life | 1 month or later after patient death
  In this exploratory outcome, bereaved caregivers will be asked to complete a 10-item validated bereaved family survey assessing their satisfaction with end-of-life care received by the patient. Domains assessed will include physical and emotional support, focus on the individual, and shared decision making. Higher scores indicate greater satisfaction with care.

CONTACTS AND LOCATIONS:
Overall Officials: Sarguni Singh, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States